CLINICAL TRIAL: NCT00428077
Title: A Multi-Center Pilot Phase II Trial of a Synthetic Tumor-Specific Breakpoint Peptide Vaccine in Patients With Chronic Myeloid Leukemia (CML) and Minimal Residual Disease
Brief Title: Vaccine Therapy in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn because there were no dramatic changes in the main endpoint, as well as low enrollment numbers. The data are not interpretable in terms of efficacy.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000526322; OHSU-HEM-05053-L; OHSU-1358
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2011-08-31 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Leukemia
Keywords: Philadelphia chromosome positive (Ph+) chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bcr-abl peptide vaccine — Patients will be vaccinated 15 times over 12 months with a vaccine comprised of native and synthetic break-point cluster region-Abelson murine leukemia(BCR-ABL) specific peptides and the immunologic adjuvants, Montanide ISA 51-VG.
Genetic: reverse transcriptase-polymerase chain reaction — A "baseline" reverse transcriptase-polymerase chain reaction(RT-PCR) transcript level of BCR-ABL will be determined after enrollment on study. This baseline will be used to measure response to the vaccine. Patients will have 3 quantitative RT-PCR tests for BCR-ABL transcript levels performed on their peripheral blood in the first month after enrolling on study. Peripheral blood samples will be drawn at approximately 1-month prior (about day -30), 2 weeks prior (about day -14), and the day of the first vaccination (day 0). Samples will be analyzed at a central lab and the three values will be averaged to determine a "baseline" circulating transcript level. During this one-month period, a peripheral blood sample will be analyzed to determine whether patients have a B3A2 or B2A2 junction.

SUMMARY:
RATIONALE: Vaccines made from a peptide may help the body build an effective immune response to kill cancer cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antileukemic effects of tumor-specific Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL) junction specific peptide vaccine, as measured by a decrease in circulating BCR-ABL transcripts by reverse-transcriptase polymerase chain reaction (RT-PCR), that persist for at least 3 months, in patients with chronic phase chronic myelogenous leukemia.
* Determine the percentage of patients treated with this vaccine who become RT-PCR-negative for BCR-ABL transcripts.
* Compare response in patients with B3A2 junctions vs B2A2 junctions when treated with this vaccine.
* Determine the immunologic response over 1 year in patients treated with this vaccine.
* Correlate response with specific HLA types in these patients.
* Determine the safety of this vaccine in these patients.

OUTLINE: This is a pilot, multicenter study.

Patients receive BCR-ABL junction-specific peptide vaccine subcutaneously in weeks 2, 4, 6, 8, and 11 and then once monthly for 10 months.

BCR-ABL transcript levels are assessed by quantitative reverse-transcriptase polymerase chain reaction at baseline, weeks 2, 4, and 6, every 3 months during treatment, and then 2 weeks after completion of study treatment.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Philadelphia chromosome-positive or BCR-ABL-positive chronic phase chronic myelogenous leukemia (CML)

  * In complete cytogenetic remission confirmed by 2 bone marrows ≥ 1 month apart
  * Minimal residual disease
* Detectable BCR-ABL transcript levels obtained < 6 months apart AND ≤ 0.5-log lower than the lowest value obtained within the past 6 months

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Bilirubin < 2 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* ALT and AST < 2.5 times ULN

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* No major surgery within the past 4 weeks
* No prior chemotherapy
* No prior immunosuppressive therapy
* No prior corticosteroids
* No prior stem cell transplantation
* No radiotherapy within the past 4 weeks
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Deininger, MD, PhD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from patient database in medical clinic.
Groups:
- Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL): Patients will be vaccinated 15 times over 12 months with a vaccine comprised of native and synthetic BCR-ABL (break-point cluster region-Abelson murine leukemia) specific peptides and the immunologic adjuvants, Montanide ISA 51-VG.
Period: Overall Study
Arm/Group | Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 59.75 (3.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One-log Decrease in Circulation Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL) Transcripts That Persists for at Least Three Months During the 1-year Treatment Period.
Description: One-log decrease in circulating BCR-ABL transcripts (RT-PCR) that persists for at least three months during the 1-year treatment period.
Time Frame: Every 3 months for the duration of the 1-year treatment period. .
Population: Per protocol.
Measure: Number; unit: Participants
Groups:
- Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL): Patients with Philadelphia Chromosome (Ph+) or Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL),positive Chronic Myeloid Leukemia(CML), in cytogenetic remission, with minimal residual disease.
Arm/Group | Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL)
Number analyzed (Participants) | 4
Participants | 4 [10 to 30]

2. Primary Outcome: Percentage of Patients Who Become RT-PCR-negative for BCR-ABL Transcripts
Time Frame: 12-24 Months
Reporting Status: Not Posted

3. Primary Outcome: Comparison of Response in Patients With B3A2 Junctions vs B2A2 Junctions
Time Frame: 12-24 Months
Reporting Status: Not Posted

4. Primary Outcome: Immunologic Response Over 1 Year
Time Frame: 12 months
Reporting Status: Not Posted

5. Primary Outcome: Correlation of Response With Specific HLA Types
Time Frame: 12-24 Months
Reporting Status: Not Posted

6. Secondary Outcome: Safety of a Vaccine Containing Native and Synthetic Chronic Myeloid Leukemia (CML) Peptides Over 1 Year Treatment.
Time Frame: Weeks 2, 4, 6, 9, and monthly thereafter up to 2 years.
Reporting Status: Not Posted
Measure: Number; unit: participants

ADVERSE EVENTS:
Time Frame: Adverse events were measured during entire 12 month period subjects received study drug.
Arm/Group | Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL)
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL) (N=4)
Acute Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1) — In one patient a grade 3 GI AE (acute gastroenteritis) occurred and led to hospitalization. This event was felt to be unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breakpoint Cluster Region-Abelson Murine Leukemia(BCR-ABL) (N=4)
Injection site induration (Skin and subcutaneous tissue disorders) | 4 (4) — All patients developed grade 1-2 injections site indurations, which slowly resolved over several months.
Fatigue (General disorders) | 3 — Patients experienced grade 1-2 fatigue in association with the injection of GM-CSF. This is an established side effect of the agent.
Cataracts (Eye disorders) | 1 (1) — One patient was diagnosed with grade 2 cataracts while on study. Given that this is common in the patient's age group, it is unlikely to be related to study medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No